CLINICAL TRIAL: NCT04114422
Title: A Feasibility Study for a Randomized Controlled Trial of a Seven-day Preoperative Exercise Training Program in People With Abdominal Cancer
Brief Title: A Seven-day Preoperative Exercise Training Program in People With Abdominal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Adriana Claudia Lunardi, Principal Investigator, Universidade Cidade de Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNICID/ 13004319.0.3001.5463
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Abdominal Cancer
Keywords: cancer; surgery; exercise training; physical therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Seven-day preoperative exercise training program (Experimental): All patients will undergo to seven-day preoperative exercise training program that includes aerobic and resistance exercises
  Interventions: Other: Seven-day preoperative exercise training program

INTERVENTIONS:
Other: Seven-day preoperative exercise training program — The preoperative exercise training program will be supervised by a physiotherapist and will comprise aerobic exercise on a treadmill as well as strengthening exercises for the upper and lower limbs. The protocol will include 7 daily sessions of 60 minutes in duration. The treadmill exercise will start with a 5-minute warm-up and will progress to 30 minutes of exercise with a speed corresponding to 70% of the maximum speed reached in the incremental shuttle walk test. It will finish with a 5-minute cool down period. Participants will also perform three strengthening exercises for the lower limbs (hip flexion, knee flexion and extension) and three for the upper limbs (shoulder flexion, elbow flexion and extension). The initial strengthening exercises intensity will be set at 60% of 1RM and will be progressively increased. Patients will perform 3 sets of 8 to 12 repetitions for each exercise.

SUMMARY:
Background: Preoperative exercise training programs of long duration, that delay surgical resection of tumors, may not be feasible in the treatment of malignant disease. In people with lung cancer, improvements in postoperative outcomes have been demonstrated with short duration (i.e. up to seven days) preoperative exercise training programs. However, the feasibility of short duration preoperative exercise training programs in people with abdominal cancer has not been investigated.

Objective: In people undergoing surgical resection for abdominal cancer, to investigate the effects of a seven-day preoperative exercise training program on preoperative exercise capacity and peripheral muscle strength as well as adherence rates, adverse events and subjective perception of satisfaction and discomfort of participants to the preoperative treatment.

Design: A feasibility study. Setting: Participants will be recruited from the surgical ward of a public hospital in São Paulo, Brazil.

Participants: 22 inpatients over 18 years old, awaiting surgical resection for colorectal, esophageal, gastric, hepatic or pancreatic cancer.

Intervention: The participants will undergo a seven-day, inpatient preoperative exercise training program that includes aerobic and resistance exercises.

Measurements: preoperative exercise capacity, peripheral muscle strength, adherence rates (consent rates, recruitment rates, completion rates and adherence), adverse events, the reasons for ineligibility and the reasons for declining participation and the subjective perception of satisfaction and discomfort of the participants to the preoperative treatment.

DETAILED DESCRIPTION:
Patients from the General Surgery ward at the Institute of Medical Assistance to Employed of São Paulo, Brazil, will be identified. Potential participants will be provided with a participant information sheet and, for those willing to participate in the study, a written informed consent will be obtained. The reasons for ineligibility and the reasons for declining participation will be recorded. Both before and following the intervention period, participants will complete assessments over a single day. Measures will be collected of: anthropometric and clinical data, preoperative exercise capacity and peripheral muscle strength. Following the completion of the intervention period, adherence rates (consent rates, recruitment rates, completion rates and adherence), adverse events and the subjective perception of satisfaction and discomfort of the participants to the preoperative treatment will also be recorded. The preoperative exercise training program will be supervised by a physiotherapist and will comprise aerobic exercise on a treadmill as well as strengthening exercises for the upper and lower limbs. The protocol will include 7 daily sessions of 60 minutes in duration. The first session will occur the day following the initial assessments. The treadmill exercise will start with a 5-minute warm-up and will progress to 30 minutes of exercise with a speed corresponding to 70% of the maximum speed reached in the incremental shuttle walk test. It will finish with a 5-minute cool down period. The intensity goal for the treadmill exercise will be to generate a rate of perceived exertion (on the dyspnea scale that ranges between 6 and 20) between 12 and 16. Exercise intensity (i.e. walking speed) will be progressively increased if the participant is able to walk for 30 minutes continuously reporting tolerable symptoms (dyspnea<12 points). Participants will also perform three strengthening exercises for the lower limbs (hip flexion, knee flexion and extension) and three for the upper limbs (shoulder flexion, elbow flexion and extension). The initial strengthening exercises intensity will be set at 60% of 1 Maximum Repetition and will be progressively increased. Patients will perform 3 sets of 8 to 12 repetitions for each exercise. The increment in exercise intensity will occur when the participant is able to perform at least 2 sets of 15 repetitions reporting tolerable symptoms (i.e. dyspnea<12 points).

Heart rate, peripheral oxygen saturation, dyspnea and blood pressure will be measured before, during (if needed; i.e. if symptoms are reported) and after each exercise training session. The session may be interrupted at any time if the patient presents major symptoms of dizziness, nausea or intolerable dyspnea/fatigue. Following surgery, all participants will receive routine physiotherapy care by the Physiotherapy team of the Institute of Medical Assistance to Employed of São Paulo

ELIGIBILITY:
Inclusion Criteria:

* Patients are over 18 years of age;
* Diagnosis of colorectal, esophageal, gastric, hepatic or pancreatic cancer;
* Hospitalization at the Institute of Medical Assistance to Employed of São Paulo, awaiting major abdominal resection (i.e. ≥ 180 minutes in duration) with a curative intent;
* Being scheduled to be hospitalized for at least 11 days before surgical resection;
* Without previous treatment for their malignancy.

Exclusion Criteria:

* musculoskeletal conditions or cognitive impairment that interferes with the proposed assessments and intervention;
* serious diseases such as heart disease (moderate to severe pulmonary aortic stenosis, decompensated heart failure, advanced cardiac arrhythmias, myocarditis, unstable coronary insufficiency, for example), lung disease (obstructive pulmonary disease and / or decompensated asthma, for example), decompensated diabetes and decompensated systemic arterial hypertension
* participation in pulmonary rehabilitation or engagement in regular physical activity in the previous 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Preoperative exercise capacity | One day before and one day after seven-day preoperative exercise training program
  Preoperative exercise capacity will be assessed via the incremental shuttle walk test. The test consists of walking on a 10 m course, around two cones positioned 9 m from each other and 0.5 m before of each end. The speed is dictated by audio signals recorded on a cell phone and progressively increases every minute. Participants will be instructed to follow the speed dictated by the audio signals until they are no longer able to keep up with the speed. The test will be terminated by either the participant, due to symptoms that make it impossible to maintain the required speed, or the assessor, if the participant fails to complete two shuttles in the time given or if the assessor judges the participant is unable to continue (e.g. peripheral oxygen saturation below 80%).

SECONDARY OUTCOMES:
Peripheral muscle strength | One day before and one day after seven-day preoperative exercise training program
  Peripheral muscle strength will be assessed by a maximum repetition test (1RM). First, the participant will perform 3-5 minutes of light activities involving the muscle groups to be tested (hip flexors, knee flexors and extensors, elbow flexors and extensors). After one minute of light stretching, the patient will perform a warm up that includes eight repetitions at 50% of 1RM perceived, followed by three repetitions at 70% of 1RM perceived. The 1RM test will be conducted following a 5 minutes interval. Additional weights will be added as needed, and three to five attempts will be performed. The maximum weight lifted in a single movement will be recorded.
Adherence rates | During 7 intervention days
  Adherence rates will be assessed by: consent rates (proportion of patients who agreed to participate in the study relative to those who were selected); recruitment rates (proportion of participants recruited relative to those who were eligible), completion rates (proportion of participants allocated that completed the intervention) and adherence (proportion of exercise training sessions completed). The reasons for ineligibility will be recorded. Reasons for declining participation will also be recorded for each patient who refuses to participate in the study.
Adverse events | During 7 intervention days
  Adverse events (e.g. dizziness, nausea, falls, fatigue) will be systematically recorded throughout the intervention period.
Subjective perception of satisfaction and discomfort of participants to the preoperative treatment. | On the day after finishing the intervention (8th day of the protocol)
  Subjective perception of satisfaction and discomfort of participants to the preoperative treatment will be assessed, via 2 questions, on completion of the intervention period. Participants will rate their satisfaction and discomfort on a scale ranging between 0 and 10. For the question about treatment satisfaction, 0 will indicate "total dissatisfaction" and 10 "maximum satisfaction". In the question is about discomfort of treatment, 0 will indicate "no discomfort" and 10 "maximum discomfort".

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Lunardi, PhD, Study Director — Universidade Cidade de São Paulo
Locations (1):
- Instituto de Assistência Médica ao Servidor Público Estadual, São Paulo, Brazil